CLINICAL TRIAL: NCT06322953
Title: A Randomised Trial of Timing to Restart Direct Oral Anticoagulants After Traumatic Intracranial Haemorrhage
Brief Title: Timing to Restart Direct Oral Anticoagulants After Traumatic Intracranial Haemorrhage
Acronym: RESTARTtlCrH
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Walton Centre NHS Foundation Trust (Other)
Collaborators: University of Liverpool (Other); National Institute for Health Research, United Kingdom (Other Government); University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG442-21
Record Dates: First submitted 2024-02-26; First posted 2024-03-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Traumatic Intracranial Haemorrhage
Keywords: Direct Oral Anticoagulants; Randomised Trial
MeSH Terms: conditions — Intracranial Hemorrhage, Traumatic | interventions — Factor Xa Inhibitors; apixaban; Dabigatran; edoxaban; Rivaroxaban

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Start/Restart DOAC at 1 week (Active Comparator): Participants will be restarted/started on DOAC 1 week post traumatic intracranial hemorrhage (tICrH).
  Interventions: Drug: Direct-Acting Oral Anticoagulants (used as per local standard practice)
- Start/Restart DOAC at 4 weeks (Active Comparator): Participants will be restarted/started on DOAC 4 weeks post traumatic intracranial hemorrhage (tICrH).
  Interventions: Drug: Direct-Acting Oral Anticoagulants (used as per local standard practice)

INTERVENTIONS:
Drug: Direct-Acting Oral Anticoagulants (used as per local standard practice) — Direct-acting oral anticoagulants to be prescribed as per local standard practice at either 1 or 4 weeks.
  Other Names: Apixaban; Dabigatran Etexilate Mesilate; Edoxaban; Rivaroxaban

SUMMARY:
Older people falling from a standing height is the most common cause of hospital admission for head injury. Up to 1 in 3 patients admitted are taking a tablet medication which thins the blood, known as an oral anticoagulant. This type of medication can increase the likelihood of bleeding in the brain. Many patients are taking oral anticoagulation due to having an irregular heartbeat (called atrial fibrillation) or because of having a previous stroke or blood clots. When a scan shows blood in the brain, oral anticoagulation is nearly always stopped. However, this leaves the question of when it is safe to restart them. The risk of making the bleeding in the brain worse must be balanced against the risk of having a stroke or blood clots. There is no clear evidence on the safest time to restart oral anticoagulation, but most neurosurgeons advise restarting them 1-4 weeks after head injury. The number of people who have a bleed on their brain after a head injury is increasing and further brain bleeding or a stroke can have a serious effect on patients' lives and their on-going healthcare needs. Public and patient groups have highlighted that many patients want to stop taking oral anticoagulation after a bleed but they may be unaware of the vital importance of restarting this medication to prevent strokes and blood clots. The most popular oral anticoagulation prescribed has changed in recent years from warfarin to newer medications called Direct Oral Anti-Coagulants (DOACs).

This trial will recruit 1084 people who are admitted to hospital with a bleed on the brain caused by a head injury who were taking oral anticoagulation before their head injury and have been prescribed a Direct Oral Anti-Coagulant (DOAC) for previously diagnosed medical condition. Patients on other Oral Anti-Coagulants, such as Warfarin may also be able to take part. The main purpose of the trial is to determine when is most beneficial time for people to start or restart a DOAC after their head injury. People will be asked to start the medication either 1 week or 4 weeks after their head injury. They will be then followed closely for 12 weeks and any major bleeding events or a blood clots (thrombotic events) such as a stroke or heart attack will be recorded. The study will also look at the person's overall quality of life, how they recover physically, the number of people who die, the costs of the treatment, and the attitudes of people and their caregivers to starting or restarting a DOAC.

DETAILED DESCRIPTION:
Head injury in older patients is becoming increasingly common. The 2017 England and Wales trauma network review reports an older person falling from standing height as the commonest type of major trauma, and most frequently results in injury to the head. By 2050, 1 in 6 people will be aged over 65, and with approximately 30% of older adults falling each year, the incidence of head injury will rise. In conjunction, there is a high prevalence of oral anticoagulant (OAC) use in this older population, driven by increased incidence of atrial fibrillation (AF), the commonest heart rhythm disorder, which is related to aging. It increases the risk of stroke 5-fold and should be considered for treatment with oral anticoagulants OACs depending on risk factor assessment by the CHA2DS2VASc (C - Congestive heart failure (1 point) H - Hypertension (1 point) A2 - Age ≥75 years (2 points) D - Diabetes mellitus (1 point) S2 - Prior Stroke or transient ischemic attack (2 points) V - Vascular disease (e.g., peripheral artery disease, myocardial infarction, aortic plaque) (1 point) A - Age 65-74 years (1 point) Sc - Female sex category (1 point) score). OAC prescribing for such patients has more than doubled in the United Kingdom (UK) since 20008 and between 20-35% of older patients admitted with head injury causing intracranial haemorrhage (tICrH), are taking an OAC at the time of injury. Standard care dictates that OACs should be stopped in the majority of cases to reduce the risk of progressive or new ICrH. Despite a low risk of new or on-going Intracranial Hemorrhage (ICrH) 48 hours after injury, there is a reluctance from clinicians to restart OACs for fear of evoking re-bleeding. This must be balanced against the increased risk of thromboembolism in patients not taking their OAC, predisposing AF patients to increased risk of stroke, systemic thromboembolism and all-cause mortality. Currently there is no clear consensus on the optimal practice on the timing for restarting OACs post- traumatic intracranial hemorrhage (tICrH). OAC medications are traditionally divided into vitamin K antagonists (e.g., warfarin) and Direct Oral Anticoagulants (DOACs). DOAC prescribing has increased substantially over the last decade. Benefits include an immediate therapeutic effect, fixed dosing, fewer drug interactions and no monitoring when compared to warfarin. Previous meta-analyses and trials demonstrate that DOACs are at least as effective as warfarin in the prevention of stroke in AF patients, and have a lower rate of associated ICrH and mortality. DOACs (eg Apixaban, dabigatran, edoxaban and rivaroxaban) are recommended by The National Institute for Health and Care Excellence (NICE) for those over 65 with AF and a CHA2DS2VASc score of 2 or above and considered for men with AF and a CHA2DS2VASc score of 16. For those already taking a Vitamin K antagonist (VKA) (e.g., Warfarin) NICE recommends that the option of switching to a DOAC should be discussed. This study will focus on patients who are taking a DOAC or Vitamin K antagonist for AF or venous thromboembolism (VTE) at the time of tICrH which is stopped due to risk of further bleeding. Patients will then either be restarted on their DOAC, or the option of switching to a DOAC from their current Vitamin K antagonist will be discussed, as these have a superior safety profile (significantly reduced risk of haemorrhagic stroke and intracerebral haemorrhage compared to warfarin) and reflects best practice following tICrH.

Studies suggest evidence of early tICrH expansion (within 48hrs) on routine repeat imaging occurs in 10-37% of patients on OAC, indicating the need to stop OAC. This risk reduces substantially over time. A recent trial assessing patients with a major bleed on OACs, reported re-bleeding rates of 4.3% within 30 days, when excluding the first 3 days from the initial bleed. The bleeding rate was only 4.5% in those who restarted their OAC within 2 weeks, with a net benefit (Hazard ratio 0.384 combining thrombosis, bleeding and death rate) when compared to those that did not restart OAC within 2 weeks. Another study focusing on tICrH reported a 5% readmission rate for re-bleeding within 30-days in patients who did not restart their DOAC. There is a paucity of high-level data on delayed (>72hrs) haemorrhage rates after tICrH and withholding OACs results in an elevated risk of thrombotic events such as stroke, myocardial infarction (MI) and VTE. A trial of 352 patients suffering a major bleed whilst on a DOAC demonstrated that thrombotic events increase from around 4% at 1 week to 10% at 4 weeks. At 3 months, patients who have restarted OAC have fewer strokes [Hazard Ratio (HR) 0.85, 95% confidence intervals (CI) 0.43-1.68] and deaths [HR 0.5, 95% CI 0.35-0.72], despite increased bleeding [HR 1.62, 95% CI 0.95-2.75] compared to those who have not restarted OAC.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained from participant / participants' legal representative / participants' Consultee and ability to comply with the requirements of the trial
2. Adult ≥18 years with traumatic intracranial haemorrhage (tICrH) in the past 1 week who were taking oral anticoagulants (OAC) prior to admission
3. Oral anticoagulants include any DOAC or Vitamin K antagonist (VKA) (e.g. Warfarin), prescribed for atrial fibrillation (AF) or venous thromboembolism (VTE) prior to admission for tICrH
4. At high risk for thromboembolic complications (CHA2DS2VASc ≥2 in men and ≥3 in women)

Exclusion Criteria:

1. Patients whose traumatic intracranial haemorrhage is a chronic subdural haematoma
2. Patients with mechanical heart valve
3. Patients with plan to start/restart anti-platelet therapy within 12 weeks of tICrH
4. Abbreviated Injury Scale other than head with a score >3
5. Pregnancy
6. Participants with a hypersensitivity or contraindication to Direct Oral Anticoagulant (DOAC)
7. Participant with bleeding where it would be unsafe to restart DOAC at 1 week
8. Participant with clinical reason to restart DOAC before 4 weeks or complete within 12 weeks
9. Concomitant p-gp and CYP3A4 inducers/inhibitors
10. Indication to stay on VKA (Warfarin) rather than switching to DOAC (e.g. severe renal impairment)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1084 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with haemorrhagic or thrombotic event within 12 weeks following tICrH. | 12 weeks
  The total number of patients that have a haemorrhagic or thrombotic event within 12 weeks following tICrH.

SECONDARY OUTCOMES:
Time to first haemorrhagic or thrombotic event. | 12 weeks
  Time to first haemorrhagic or thrombotic event.
Time to first haemorrhagic event | 12 weeks
  Time to first haemorrhagic event
Time to first thrombotic event | 12 weeks
  Time to first thrombotic event
Time to death | 12 and 26 weeks
  Time to death
Functional outcome measured using modified Rankin Scale (mRS) | 12 and 26 weeks
  The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. The scale ranges from 0-6 with 0 being no symptoms and 6 being dead.
Functional outcome measured using Barthel Index | 12 and 26 weeks
  The barthel index is a tool to rank the patient's independence in 10 areas of daily living, such as feeding, bathing, dressing, and mobility. The total score ranges from 0-100 with 0 having no independence and 100 being totally independent.
Functional outcome measured using extended Glasgow Outcome Scale (GOS-E) | 12 and 26 weeks
  The scale runs from 0-6, running from perfect health without symptoms to death. The Extended Glasgow Coma Scale (EGCS) expands upon the traditional GCS by adding additional components to provide a more comprehensive assessment of a patient's neurological status. It consists of 8 levels with 1 being dead and 8 meaning patient has made a complete recovery.
Overall Quality of Life measured by EuroQol 5 Dimensions 5 Levels (EQ5D5L) questionnaire | 12 and 26 weeks
  The EuroQol 5 Dimensions 5 Levels (EQ5D5L) is a standardized instrument used for measuring generic health status and health-related quality of life. This system comprises five dimensions of health: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has five levels of severity, ranging from no problems to extreme problems. In addition to the descriptive system, the EQ5D5L includes a vertical visual analogue scale (VAS) where respondents rate their current health on a scale from 0 to 100, with 0 representing the worst imaginable health state and 100 representing the best imaginable health state.
Patient/caregiver attitudes to (re)starting OAC | Within the first 9 months of recruitment start
  This qualitative sub-study will explore patient and caregiver attitudes to recommencing a DOAC following tICrH. An individual semi-structured interview, lasting 30-60 minutes with a qualitative researcher will be undertaken to elicit their perceptions and beliefs about DOACs, in relation to stroke prevention and risks of recurrent ICrH. The interview will be conducted in person/remotely (depending on participant preference) within 60 days of the study approach.
Healthcare resource use | 6, 12 and 26 weeks
  A client service receipt inventory questionnaire (CSRI) will be administered to participants to collect information regarding healthcare services used. The CSRI will collect detailed data on visits to general practitioners, specialists, hospital admissions, outpatient appointments, and mental health services. Services accessed such as home care, day care, residential care, and support services for individuals with disabilities or mental health needs. Information about prescription medications and over-the-counter drugs taken. informal care provided by family members or friends, as well as other forms of support such as transportation services or assistance with daily living activities. The data collected through the CSRI will be used to quantify the costs associated with different types of services and interventions, assess the impact of services on outcomes such as quality of life or functioning, and inform decision-making in healthcare and social care policy.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine McMahon, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - University Hospitals Plymouth NHS Trust, Plymouth, Devon
  - The Walton Centre NHS Foundation Trust, Liverpool, Mersyside

IPD SHARING:
Plan to Share IPD: No
Anonymous data will be available on request following the end of the study.